CLINICAL TRIAL: NCT03590964
Title: One-stage Maxillary Sinus Elevation Using a Bone Core Containing an Implant From the Mandibular Symphysis: (A Randomized Controlled Trial)
Brief Title: One-stage Maxillary Sinus Elevation Using a Bone Core Containing an Implant From the Mandibular Symphysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed kamel hassan, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-07-05
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Atrophied Posterior Maxilla
Keywords: Implant, Bone ring, Sinus lift.

STUDY DESIGN:
Intervention Model Description: * A Randomized controlled trial.
  * Parallel group study.
  * A trial will be carried out in hospital of Oral and Maxillofacial surgery department- Faculty of Oral and Dental Medicine Cairo University
  * Equal randomization: participants with equal probabilities for intervention.
  * Positive controlled: Both groups receiving treatment.
Masking Description: Because the two interventions used in this trial are clearly different and easily recognized by the participants and investigators, neither the investigators nor participants can be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open sinus lift using chin bone graft (Active Comparator): Patients with atrophied posterior maxilla will undergo open sinus lift with chin bone graft according to standardized surgical approach.
  Interventions: Procedure: Open sinus lift using chin bone graft
- Sinus lift using bone ring containing the implant (Experimental): Patients with atrophied posterior maxilla will undergo sinus lift using bone ring containing the implant.
  Interventions: Procedure: Sinus lift using bone ring containing the implant.

INTERVENTIONS:
Procedure: Open sinus lift using chin bone graft — Patients with atrophied posterior maxilla will undergo open sinus lift with chin bone graft according to standardized surgical approach.
  Other Names: Lateral sinus approach with chin graft
  Arms: Open sinus lift using chin bone graft
Procedure: Sinus lift using bone ring containing the implant. — Patients with atrophied posterior maxilla will undergo sinus lift with chin bone ring containing the implant.
  Other Names: One stage sinus lift using bone ring
  Arms: Sinus lift using bone ring containing the implant

SUMMARY:
Two groups of patients with atrophy in posterior maxilla indicated for sinus lift.

First group will be subjected to open sinus lift with chin bone graft. Second group will be subjected to sinus floor elevation using a bone ring.

DETAILED DESCRIPTION:
Two groups of patients with atrophy in posterior maxilla indicated for sinus lift.

(A) First group will be subjected to open sinus lift with chin bone graft.

* All cases will undergo surgery under general anesthesia for sinus lift and other surgery under local anesthesia for implant placement .
* Exposure of the anterior wall of maxilla according to standardized surgical approach.
* Open sinus lift and bone graft.
* After 6 months, implant will be drilled and inserted in the recipient site according to standard protocol.
* Loading on implant after 5-6 months.

(B)Second group will be subjected to sinus floor elevation using a bone ring.

* All cases will undergo surgery under local anesthesia for implant placement in the mandibular chin and other surgery under general anesthesia for sinus lift using bone ring with the implant.
* Exposure of the mandibular chin will be done under local anesthesia using a standardized surgical approach.
* Implant will be drilled and inserted in the chin according to standard protocol.
* After 3 months, second surgery under general anesthesia to place the implant and surrounding ring in the atrophied posterior maxilla.
* The bone ring containing the implant allowed to heal for 5-6 months.

Follow up:

* Clinical evaluation will be performed at the first week post-operative.
* Three months post-operative second surgery to put the implant with surrounding ring in atrophied posterior maxilla.
* Five months post-operative to the second surgery, implant will be loaded with the final restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least a unilateral atrophied posterior maxilla indicated for open sinus lift and graft.
2. All ages and both sexes were included in this study.
3. Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
4. Patients with good general condition allowing surgical procedure under general anesthesia.
5. Patients with physical and psychological tolerance.

Exclusion Criteria:

1. Patients with high risk systemic diseases like uncontrolled diabetes. As uncontrolled diabetes has a negative impact on normal bone healing.
2. Patients with chronic sinusitis, maxillary sinus tumor or cyst. As they will affect accuracy of the procedure.
3. Patients with physical and psychological intolerance. As psychological stress will affect the immune system and patient's fitness including healing capacity. ]

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate of implant | One year post-operative.
  The estimated annual failure rate will be assessed via clinical assessment, measuring unit (Binary yes\ no)

SECONDARY OUTCOMES:
Marginal bone loss around implant | one year post operative
  Bone loss around implant will be assessed using Cone Beam Computed Tomography, measuring unit (millimeter).
Pain intensity | One month post-operative.
  Intensity of pain will be assessed using Visual analog scale (0 -10), 0 indicate no pain,10 indicate unbearable pain.
Sinus membrane perforation | During operation
  Perforation of sinus lining will be assessed clinically, (Binary yes\no).
Established bone integration | Six months post operative.
  Structural and functional integration of bone around implant will be assessed using a device with measuring unit scale of 1-100.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Y yassin, PhD., Study Director — Faculty of Oral and Dental Medicine- Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine-Cairo University., Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mahesh L, Kurtzman GM, Shukla S. Trephine core: an alternative sinus lift technique. J Oral Implantol. 2014 Jul;40 Spec No:391-6. doi: 10.1563/aaid-joi-D-14-00047. Epub 2014 Mar 12. No abstract available. PMID 24621196
- [Result] Wallace SS, Froum SJ. Effect of maxillary sinus augmentation on the survival of endosseous dental implants. A systematic review. Ann Periodontol. 2003 Dec;8(1):328-43. doi: 10.1902/annals.2003.8.1.328. PMID 14971260
- [Result] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Result] Wang PD, Klein S, Kaufman E. One-stage maxillary sinus elevation using a bone core containing a preosseointegrated implant from the mandibular symphysis. Int J Periodontics Restorative Dent. 2002 Oct;22(5):435-9. PMID 12449303